CLINICAL TRIAL: NCT06192368
Title: Acceptability, Feasibility, and Preliminary Effects of a Virtual Reality (VR) Program to Reduce Stress in Neonatal Intensive Care Unit Nurses
Brief Title: Virtual Reality Program to Reduce Stress in Neonatal Nurses
Acronym: INSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Sylvie Le May, Professor, St. Justine's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: INSPIRE
Record Dates: First submitted 2023-12-18; First posted 2024-01-05 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Virtual Reality; Stress; Stress, Work Place
Keywords: Virtual reality; Nurse; Stress; Anxiety
MeSH Terms: conditions — Occupational Stress; Anxiety Disorders | interventions — Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence of virtual reality followed by tablet game. (Other): Over a period of two weeks (weeks 1 and 2), participants randomized to this sequence will be asked to use virtual reality for 15 minutes during four break periods. These two weeks of virtual reality will be followed by a week with no exposure (week 3). In the following two weeks, participants will be asked to play a game on a tablet for 15 minutes during four break periods (weeks 4 and 5).
  Interventions: Device: INSPIRE; Device: Tablet
- Sequence of tablet game followed by virtual reality: (Other): Over a two-week period (weeks 1 and 2), participants randomized to this sequence will be asked to play a game on a tablet for 15 minutes during four break periods. These two weeks of tablet gaming will be followed by a week with no exposure (week 3). In the following two weeks, participants will be asked to use virtual reality for 15 minutes during four break periods (weeks 4 and 5).
  Interventions: Device: INSPIRE; Device: Tablet

INTERVENTIONS:
Device: INSPIRE — Virtual reality application for relaxing.
Device: Tablet — Gaming tablet

SUMMARY:
Background: In the context of neonatal care, the increasing complexity of medical interventions poses challenges to nurses, contributing to elevated workplace stress. This stress can impact the well-being of nurses and the overall quality of patient care. Despite the documented significance of workplace stress, there is a scarcity of research on effective stress management interventions for neonatal care nurses. This pilot study aims to explore the feasibility, acceptability, and preliminary effects of a virtual reality (VR) intervention on stress reduction among nurses in the neonatal intensive care unit (NICU) at CHU Sainte-Justine.

Methods: A randomized intra-subject clinical trial will be conducted, involving 30 NICU nurses and nurse assistants. Participants will act as their own controls, receiving both experimental (VR) and control (tablet gaming) interventions in a random sequence. The study will assess the feasibility of the interventions, clinical trial procedures, and participant satisfaction. Stress levels will be measured using the State-Trait Anxiety Inventory (Trait subscale), Nurse Stress Scale, Stress Numerical Rating Scale-11, and salivary alpha-amylase. Additionally, participants will provide sociodemographic information, and the study will evaluate the perceived clinical workload during intervention sessions.

Interventions: The study will employ Paperplane Therapeutics' VR program, INSPIRE, designed to offer a multisensory relaxation experience. The control intervention involves tablet gaming during breaks. Both interventions will be 15 minutes in duration, implemented over five weeks.

Results: The study aims to provide insights into the feasibility, acceptability, and preliminary effects of VR-based stress management interventions for NICU nurses. Data analysis will involve statistical comparisons of stress measures between VR and control interventions, contributing to the evidence base for implementing workplace stress reduction programs.

Conclusion: This research addresses a critical gap in the literature by investigating the potential benefits of VR interventions for stress reduction among NICU nurses. If successful, this approach could enhance workplace well-being, job satisfaction, and overall nursing care quality, leading to broader implications for stress management strategies in healthcare settings.

DETAILED DESCRIPTION:
INTRODUCTION In 2021-2022, there were 368,792 births in Canada, with 83,300 (22.5%) in Quebec (Canada). At the CHU Sainte-Justine, the neonatal intensive care unit admits 869 babies during the 2021-22 period. Out of these, 385 babies (44%) were born prematurely and 484 (56%) were admitted for perinatal issues or congenital pathologies. Some of these babies had to be hospitalized for several weeks or even months after birth.

The complexity of care for this population is well-documented and has consequences for nurses working daily in neonatal care units. Nurses in these units reportedly experience significant work-related stress from various stressors. Given the impact of stress on the performance of healthcare organizations, it becomes imperative for nursing unit managers, to implement measures to help nurses better manage and reduce stress in the workplace. In this context, the use of virtual reality (VR) has proven effective in stress reduction for caregivers by providing a relaxing experience. VR is a technology that simulates the user's presence in a virtual environment, visualized using a three-dimensional immersive screen inside a virtual reality headset.

To date, no studies have been identified proposing an intervention using VR for the stress management of caregivers during working hours.

AIMS & OBJECTIVES OF THE STUDY This pilot study aims to test and evaluate the feasibility, acceptability, and preliminary effects of a virtual reality activity on the stress of nursing staff in the neonatal unit at CHU Sainte-Justine during their breaks.

Objectives:

* Verify the feasibility of the intervention among participants.
* Evaluate the feasibility of the clinical trial.
* Verify the acceptability and satisfaction of nurses and nursing assistants regarding the use of VR.
* Evaluate the preliminary effects of the VR intervention on the stress levels of neonatal intensive care staff.
* Assess the feasibility of the clinical trial.

METHODS

DESIGN This is a crossover clinical trial with randomized sequences. Each participant will serve as their own control, receiving both an experimental treatment sequence (virtual reality) and a control treatment sequence (tablet game). The order of the sequences will be determined randomly. A period with no intervention (Wash out period) is planned between the two sequences to prevent the effect of the first sequence from influencing the second.

SETTING The study will take place in the neonatal intensive care unit at CHU Sainte-Justine, a reference center and one of the six tertiary and quaternary neonatal critical care units in Quebec, Canada.

INTERVENTIONS CONTROL TREATMENT Tablet gaming sessions where participants will be able to choose from several games installed on a tablet dedicated to the project.

EXPERIMENTAL TREATMENT Virtual reality sessions using the therapeutic virtual reality program INSPIRE.

VARIABLES AND MEASUREMENT INSTRUMENTS

STATE-TRAIT ANXIETY INVENTORY (STAI, TRAIT SUBSCALE ONLY) The State-Trait Anxiety Inventory (STAI) is a tool used to measure general and habitual anxiety. This scale distinguishes anxiety into emotional response (state subscale) and trait anxiety (trait subscale). Trait anxiety is defined as "relatively stable individual differences in the predisposition to perceive several situations as dangerous or threatening and to respond to these situations with an elevation of situational anxiety". The trait subscale consists of a total of 20 items where participants are asked to indicate, using a four-point Likert scale ("almost never" to "almost always"), how often they experience the mentioned emotional state. For statistical analyses, the scale results will be considered on a total of 80 points. The scores assigned to all 20 items will be summed.

NURSE STRESS SCALE (NSS) The Nurse Stress Scale (NSS) is a tool used to measure nursing stress. This questionnaire measures the frequency and sources of stress experienced by nurses during their work on care units. In this research, version 28 of the tool, consisting of 48 items, will be used. The questionnaire was pre-tested with a cohort of nurses and nursing assistants in the neonatology unit.

A 4-point Likert scale is used to indicate the frequency with which nurses experience stress factors, ranging from "never stressful" to "very often stressful." Nurses also have the option to respond N/A (not applicable) if they have never experienced the stressful item in the neonatal unit. For statistical analyses, the total score of this instrument will be considered. The scores assigned to all 43 items will be summed and then divided by the total number of items. A higher score indicates greater stress. The internal consistency of the NSS is very good (Cronbach's alpha 0.89).

An open-ended question at the end of the questionnaire will be added, asking, "In your opinion, are there other elements related to stress that you experience at work that have not been addressed by the scale and would be important to mention?"

STRESS NUMERICAL RATING SCALE-11 (SNRS-11) The perceived level of immediate stress will also be assessed using the Stress Numerical Rating Scale-11 (SNRS-11). This stress scale is a tool used to measure immediate perceived stress on a scale of 0 to 10.

SALIVARY ALPHA-AMYLASE Salivary alpha-amylase is a physiological measure of the psychosocial stress level of a participant. A decrease (or the same value as at T0 or slightly increased) or an increase between two measurement times indicates a reduction or an increase in the perceived stress level.

SOCIODEMOGRAPHIC AND CONTEXTUAL DATA A sociodemographic questionnaire will be completed by the nurses before their first gaming session. This questionnaire will be useful for describing the sample.

INTERVENTION ACCEPTABILITY AND PARTICIPANT SATISFACTION After their final gaming session, participants will be invited to complete a questionnaire regarding their appreciation of virtual reality, the ease of technology use, the support or obstacles they encountered during their participation, and their overall satisfaction with the intervention.

ANALYSES The analyses will be performed using the statistical analysis software SPSS 29th edition, IBM, Armonk, NY, USA. Descriptive statistics will be used to present sociodemographic and contextual data as well as the satisfaction levels of healthcare professionals. To control for intra- and inter-subject variability, the investigators will use RM-Anova for comparison between different stress measurement times.

The investigators will proceed with a subgroup analysis for the number of years of experience in intensive care, as well as by job title. The investigators will use a significance threshold of 0.05, but considering that this project is a pilot study, they do not aim to verify the effectiveness of VR.

ETHICAL CONSIDERATIONS This project was approved by the Research Ethics Board (REB) of CHU Sainte-Justine in Montreal, Canada.

ELIGIBILITY:
Inclusion Criteria:

- Nurses and nursing assistants holding a position or assigned to the neonatology intensive care unit

Exclusion Criteria:

* Epilepsy history
* Recent eye surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | Measured at baseline T0
  State-Trait Anxiety Inventory allow to measure general anxiety, likert scale (4 points)
Nurse Stress Scale (NSS) | Measured at Baseline (T0) and two weeks after (T7)
  Nurse Stress Scale allow to measure hospital related stress, likert scale (4 points)
Stress Numerical Rating Scale-11 (SNRS-11) | Before and after all the interventions (T0, 20 minutes after intervention-T1, at Day-2 (T2), 20 minutes after intervention-T3, at Day 4 (T4), 20 minutes after intervention-T5, at Day 6 (T6), 20 after minutes intervention-T7)
  0-10 scale to measure immediate stress
Salivary Alpha-amylase (SAA) | Before the first intervention (T0) and two weeks after (T7)
  Physiological measure for psychosocial stress.

CONTACTS AND LOCATIONS:
Locations (1):
- St.Justine's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen S, Mintz-Binder R, Sweatt L, Song H. Building nurse resilience in the workplace. Appl Nurs Res. 2021 Jun;59:151433. doi: 10.1016/j.apnr.2021.151433. Epub 2021 Apr 14. PMID 33947518
- [Background] Bekelepi N, Martin P. Support interventions for nurses working in acute psychiatric units: A systematic review. Health SA. 2022 Apr 29;27:1811. doi: 10.4102/hsag.v27i0.1811. eCollection 2022. PMID 35548058
- [Background] Beverly E, Hommema L, Coates K, Duncan G, Gable B, Gutman T, Love M, Love C, Pershing M, Stevens N. A tranquil virtual reality experience to reduce subjective stress among COVID-19 frontline healthcare workers. PLoS One. 2022 Feb 9;17(2):e0262703. doi: 10.1371/journal.pone.0262703. eCollection 2022. PMID 35139092
- [Background] Bodet-Contentin L, Letourneur M, Ehrmann S. Virtual reality during work breaks to reduce fatigue of intensive unit caregivers: A crossover, pilot, randomised trial. Aust Crit Care. 2023 May;36(3):345-349. doi: 10.1016/j.aucc.2022.01.009. Epub 2022 Mar 1. PMID 35246356
- [Background] Canada, S. (2022). Estimations des composantes de l'accroissement démographique, annuelles https://doi.org/https://doi.org/10.25318/1710000801-fra
- [Background] Crompton, S. (2011). Qu'est-ce qui stresse les stressés? Principales sources de stress des travailleurs https://www150.statcan.gc.ca/n1/fr/pub/11-008-x/2011002/article/11562-fra.pdf?st=CL4LBGSE
- [Background] Currie K, Gupta BV, Shivanand I, Desai A, Bhatt S, Tunuguntla HS, Verma S. Reductions in anxiety, depression and insomnia in health care workers using a non-pharmaceutical intervention. Front Psychiatry. 2022 Sep 6;13:983165. doi: 10.3389/fpsyt.2022.983165. eCollection 2022. PMID 36147990
- [Background] Dyrbye LN, Shanafelt TD, Johnson PO, Johnson LA, Satele D, West CP. A cross-sectional study exploring the relationship between burnout, absenteeism, and job performance among American nurses. BMC Nurs. 2019 Nov 21;18:57. doi: 10.1186/s12912-019-0382-7. eCollection 2019. PMID 31768129
- [Background] Favrod C, Jan du Chene L, Martin Soelch C, Garthus-Niegel S, Tolsa JF, Legault F, Briet V, Horsch A. Mental Health Symptoms and Work-Related Stressors in Hospital Midwives and NICU Nurses: A Mixed Methods Study. Front Psychiatry. 2018 Aug 20;9:364. doi: 10.3389/fpsyt.2018.00364. eCollection 2018. PMID 30177890
- [Background] Fiske E. Nurse Stressors and Satisfiers in the NICU. Adv Neonatal Care. 2018 Aug;18(4):276-284. doi: 10.1097/ANC.0000000000000514. PMID 29933342
- [Background] French SE, Lenton R, Walters V, Eyles J. An empirical evaluation of an expanded Nursing Stress Scale. J Nurs Meas. 2000 Fall-Winter;8(2):161-78. PMID 11227582
- [Background] Gauthier, J., & Bouchard, S. (1993). Adaptation canadienne-française de la forme révisée du State-Trait Anxiety Inventory de Spielberger. Canadian Journal of Behavioural Science/Revue canadienne des sciences du comportement, 25(4), 559.
- [Background] Gray-Toft, P., & Anderson, J. G. (1981, 1981/03/01). The Nursing Stress Scale: Development of an instrument. Journal of behavioral assessment, 3(1), 11-23. https://doi.org/10.1007/BF01321348
- [Background] Hannan KE, Bourque SL, Palmer C, Tong S, Hwang SS. Prevalence and Predictors of Medical Complexity in a National Sample of VLBW Infants. Hosp Pediatr. 2021 May;11(5):525-535. doi: 10.1542/hpeds.2020-004945. PMID 33906959
- [Background] Haugland WA, Crenshaw JT, Gilder RE. Implementing a Resilience Bundle for Emergency Nurses: An Evidence-Based Practice Project. J Emerg Nurs. 2023 Jan;49(1):40-49. doi: 10.1016/j.jen.2022.08.009. Epub 2022 Sep 30. PMID 36184334
- [Background] Hevezi JA. Evaluation of a Meditation Intervention to Reduce the Effects of Stressors Associated With Compassion Fatigue Among Nurses. J Holist Nurs. 2016 Dec;34(4):343-350. doi: 10.1177/0898010115615981. Epub 2015 Nov 23. PMID 26598000
- [Background] Jung SE, Ha DJ, Park JH, Lee B, Kim MS, Sim KL, Choi YH, Kwon CY. The Effectiveness and Safety of Mind-Body Modalities for Mental Health of Nurses in Hospital Setting: A Systematic Review. Int J Environ Res Public Health. 2021 Aug 23;18(16):8855. doi: 10.3390/ijerph18168855. PMID 34444604
- [Background] Kwon CY, Lee B. Systematic Review of Mind-Body Modalities to Manage the Mental Health of Healthcare Workers during the COVID-19 Era. Healthcare (Basel). 2022 Jun 1;10(6):1027. doi: 10.3390/healthcare10061027. PMID 35742076
- [Background] LiaBraaten BM, Linneman N, Czarnecki ML, Davies WH, Zhang L, Simpson PM, Jastrowski Mano KE, Weisman SJ, Hainsworth KR. Stress Numerical Rating Scale-11: Validation in Pediatric Inpatient and Outpatient Pain Settings. Pain Manag Nurs. 2023 Aug;24(4):e7-e12. doi: 10.1016/j.pmn.2023.03.008. Epub 2023 Apr 12. PMID 37059666
- [Background] Linares-Chamorro M, Domenech-Oller N, Jerez-Roig J, Pique-Buisan J. Immersive Therapy for Improving Anxiety in Health Professionals of a Regional Hospital during the COVID-19 Pandemic: A Quasi-Experimental Pilot Study. Int J Environ Res Public Health. 2022 Aug 9;19(16):9793. doi: 10.3390/ijerph19169793. PMID 36011433
- [Background] Lord-Gauthier J, de Montigny F, Bouchard S. Le stress au travail. Savoir y faire face. Perspect Infirm. 2016 Nov-Dec;13(5):21-25. No abstract available. French. PMID 29381275
- [Background] Martin P, Lizarondo L, Kumar S, Snowdon D. Impact of clinical supervision on healthcare organisational outcomes: A mixed methods systematic review. PLoS One. 2021 Nov 19;16(11):e0260156. doi: 10.1371/journal.pone.0260156. eCollection 2021. PMID 34797897
- [Background] Michael SH, Villarreal PM, Ferguson MF, Wiler JL, Zane RD, Flarity K. Virtual Reality-Based Resilience Programs: Feasibility and Implementation for Inpatient Oncology Nurses. Clin J Oncol Nurs. 2019 Dec 1;23(6):664-667. doi: 10.1188/19.CJON.664-667. PMID 31730607
- [Background] Mintz-Binder R, Andersen S, Sweatt L, Song H. Exploring Strategies to Build Resiliency in Nurses During Work Hours. J Nurs Adm. 2021 Apr 1;51(4):185-191. doi: 10.1097/NNA.0000000000000996. PMID 33734177
- [Background] Monroe C, Loresto F, Horton-Deutsch S, Kleiner C, Eron K, Varney R, Grimm S. The value of intentional self-care practices: The effects of mindfulness on improving job satisfaction, teamwork, and workplace environments. Arch Psychiatr Nurs. 2021 Apr;35(2):189-194. doi: 10.1016/j.apnu.2020.10.003. Epub 2020 Oct 13. PMID 33781399
- [Background] Muir KJ, Webb-Jones J, Farish N, Barker K, Miller-Davis C, Galloway S. "Room to Reflect": A Pilot Workplace Resiliency Intervention for Nurses. Int J Environ Res Public Health. 2022 Jun 14;19(12):7272. doi: 10.3390/ijerph19127272. PMID 35742534
- [Background] Murthy K, Dykes FD, Padula MA, Pallotto EK, Reber KM, Durand DJ, Short BL, Asselin JM, Zaniletti I, Evans JR. The Children's Hospitals Neonatal Database: an overview of patient complexity, outcomes and variation in care. J Perinatol. 2014 Aug;34(8):582-6. doi: 10.1038/jp.2014.26. Epub 2014 Mar 6. PMID 24603454
- [Background] Nijland JWHM, Veling W, Lestestuiver BP, Van Driel CMG. Virtual Reality Relaxation for Reducing Perceived Stress of Intensive Care Nurses During the COVID-19 Pandemic. Front Psychol. 2021 Sep 29;12:706527. doi: 10.3389/fpsyg.2021.706527. eCollection 2021. PMID 34659021
- [Background] Nowrouzi B, Giddens E, Gohar B, Schoenenberger S, Bautista MC, Casole J. The quality of work life of registered nurses in Canada and the United States: a comprehensive literature review. Int J Occup Environ Health. 2016 Oct;22(4):341-358. doi: 10.1080/10773525.2016.1241920. Epub 2016 Oct 13. PMID 27734769
- [Background] Park JH, Jung SE, Ha DJ, Lee B, Kim MS, Sim KL, Choi YH, Kwon CY. The effectiveness of e-healthcare interventions for mental health of nurses: A PRISMA-compliant systematic review of randomized controlled trials. Medicine (Baltimore). 2022 Jun 24;101(25):e29125. doi: 10.1097/MD.0000000000029125. PMID 35758346
- [Background] Penque S. Mindfulness to promote nurses' well-being. Nurs Manage. 2019 May;50(5):38-44. doi: 10.1097/01.NUMA.0000557621.42684.c4. PMID 30985526
- [Background] Rochefort CM, Clarke SP. Nurses' work environments, care rationing, job outcomes, and quality of care on neonatal units. J Adv Nurs. 2010 Oct;66(10):2213-24. doi: 10.1111/j.1365-2648.2010.05376.x. Epub 2010 Jul 2. PMID 20626479
- [Background] Rodwell J, Noblet A, Demir D, Steane P. Supervisors are central to work characteristics affecting nurse outcomes. J Nurs Scholarsh. 2009;41(3):310-9. doi: 10.1111/j.1547-5069.2009.01285.x. PMID 19723280
- [Background] Rogers, E. E., Hintz, S. R., & Gould, J. B. (2019). Quality improvement in neonatal care: Does it work for the very preterm infant? . Seminars in Perinatology, 43(6)(151156). https://www.sciencedirect.com/science/article/abs/pii/S0146000519300319
- [Background] Shepley, M. M., Harris, D. D., & White, R. (2008, 2008/03/01). Open-Bay and Single-Family Room Neonatal Intensive Care Units: Caregiver Satisfaction and Stress. Environment and Behavior, 40(2), 249-268. https://doi.org/10.1177/0013916507311551
- [Background] Stemmer R, Bassi E, Ezra S, Harvey C, Jojo N, Meyer G, Ozsaban A, Paterson C, Shifaza F, Turner MB, Bail K. A systematic review: Unfinished nursing care and the impact on the nurse outcomes of job satisfaction, burnout, intention-to-leave and turnover. J Adv Nurs. 2022 Aug;78(8):2290-2303. doi: 10.1111/jan.15286. Epub 2022 May 9. PMID 35533090
- [Background] Thacker K, Haas Stavarski D, Brancato V, Flay C, Greenawald D. CE: Original Research: An Investigation into the Health-Promoting Lifestyle Practices of RNs. Am J Nurs. 2016 Apr;116(4):24-30; quiz 31. doi: 10.1097/01.NAJ.0000482141.42919.b7. PMID 26974744
- [Background] Thomas AO, Bakas T, Miller E, Johnson K, Tubbs-Cooley HL. Burnout and Turnover among NICU Nurses. MCN Am J Matern Child Nurs. 2022 Jan-Feb 01;47(1):33-39. doi: 10.1097/NMC.0000000000000780. PMID 34860785
- [Background] Tucker SJ, Weymiller AJ, Cutshall SM, Rhudy LM, Lohse CM. Stress ratings and health promotion practices among RNs: a case for action. J Nurs Adm. 2012 May;42(5):282-92. doi: 10.1097/NNA.0b013e318253585f. PMID 22525292
- [Background] Vahedian-Azimi A, Hajiesmaeili M, Kangasniemi M, Fornes-Vives J, Hunsucker RL, Rahimibashar F, Pourhoseingholi MA, Farrokhvar L, Miller AC. Effects of Stress on Critical Care Nurses: A National Cross-Sectional Study. J Intensive Care Med. 2019 Apr;34(4):311-322. doi: 10.1177/0885066617696853. Epub 2017 Mar 10. PMID 29277137
- [Background] Walden M, Janssen DW, Lovenstein A. What Keeps Neonatal Nurses Up at Night and What Gets Them Up in the Morning? Adv Neonatal Care. 2020 Dec;20(6):E102-E110. doi: 10.1097/ANC.0000000000000723. PMID 32118649